CLINICAL TRIAL: NCT04204876
Title: Longitudinal Imaging in Patients With Large Vessel Vasculitis to Predict Further Disease Course
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Swiss Foundation for the Study of Muscular Diseases (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2019-02161; me18Daikeler
Record Dates: First submitted 2019-12-17; First posted 2019-12-19 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Giant Cell Arteritis; Large Vessel Giant Cell Arteriitis
Keywords: magnet resonance imaging (MRI); Positron emission tomography/computer tomography (PET/CT); GCA relapse
MeSH Terms: conditions — Giant Cell Arteritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- patients with GCA: All patients presenting with a new diagnosis of LV-GCA and all patients already treated for LV-GCA and planned for treatment termination
  Interventions: Diagnostic Test: Magnet Resonance Imaging (MRI); Diagnostic Test: PET/CT analysis

INTERVENTIONS:
Diagnostic Test: Magnet Resonance Imaging (MRI) — MRI with and without Gadolinium contrast agent for the following vessels: thoracic aorta (ascending, arch, descending arch, left and right common carotic, subclavian, and vertebral artery)
Diagnostic Test: PET/CT analysis — Standard value uptake measurement (SUV) based on quantitative score normalized to liver (SUV vessel max/liver mean) at the following vessel regions: Carotid artery: common, internal, external; Subclavian artery; Axillary artery; Vertebral artery; Thoracic Aorta; Abdominal Aorta; Common femoral artery; Deep femoral artery; Popliteal artery

SUMMARY:
Longitudinal imaging in patients with large vessel vasculitis to predict further disease course

DETAILED DESCRIPTION:
This explorative longitudinal prospective observational study is to explore different aspects of vessel wall characteristics as detected by magnet resonance imaging (MRI) techniques and positron emission tomography/computer tomography (PET/CT) in patients with large vessel giant cell Arteriitis (LV-GCA) for their usefulness as predictive factor for future giant cell arteritis (GCA) relapse. It analyses parameters in PET/CT and MRI in patients with GCA at treatment stop which correlate with GCA relapse within the first 6 months after treatment stop.

Patients included in the established local GCA database (BARK) will be screened for eligibility. Aortal imaging is performed during routine care according to established guidelines at diagnosis and during Follow Up at least every two years and before treatment stop.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of GCA and having a diagnosis of LV-GCA confirmed by imaging (PET/CT)
* Informed consent to the local GCA cohort BARK
* Followed for GCA treatment in the outpatient department.

Exclusion Criteria:

* Known hypersensitivity or allergy to Gadolinium (Gd)-based MRI contrast agents.
* Patients with cardiac pacemakers, intra cranial clips, metallic foreign bodies or other not MR-compatible implants (e.g. pumps etc.).
* Renal failure or severely impaired kidney function (eGFR < 30 ml/min /1,73 m2)
* Epilepsy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients presenting with a new diagnosis of LV-GCA and all patients already treated for LV-GCA and planned for treatment termination at the University Hospital Basel.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-05-28 (Actual); Primary Completion 2023-08-05 (Actual); Study Completion 2023-08-05 (Actual)

PRIMARY OUTCOMES:
Change in mural thickening at MRI analysis | at time of diagnosis of GCA and before treatment stop (in order 52 weeks after treatment start)
  0 = no mural thickening (maximal vessel wall thickness <2 mm for aorta, <1mm for its branches)
  1. = mural thickening (2-3 mm for aorta, 1-2 mm for its branches);
  2. = strong thickening (>3 mm for aorta, >2mm for its branches)

SECONDARY OUTCOMES:
Change in late mural enhancement (subjective grading) at MRI analysis | at time of diagnosis of GCA and before treatment stop (in order 52 weeks after treatment start)
  0= no mural enhancement;
  1. slight mural enhancement;
  2. strong mural enhancement and/or perivascular enhancement
Change in mural edema (subjective grading) at MRI analysis | at time of diagnosis of GCA and before treatment stop (in order 52 weeks after treatment start)
  0= no mural edema;
  1. slight mural edema;
  2. strong mural edema
Change in dynamic contrast agent uptake in Golden Angle Radial Sparse Parallel MRI (GRASP MRI) | at time of diagnosis of GCA and before treatment stop (in order 52 weeks after treatment start)
  Dynamic contrast agent uptake in GRASP will be assessed in areas with wall thickening (grade 1 or 2 as defined above)
Change in Apparent Diffusion Coefficient (ADC) as assessed with DW-MRI in absolute numbers (in mm2/s) | at time of diagnosis of GCA and before treatment stop (in order 52 weeks after treatment start)
  Apparent Diffusion Coefficient (ADC) as assessed with DW-MRI in absolute numbers (in mm2/s)
Change in Standard value uptake measurement (SUV) based on quantitative score normalized to liver (SUV vessel max/liver mean) at PET/CT analysis | at time of diagnosis of GCA and before treatment stop (in order 52 weeks after treatment start)
  Standard value uptake measurement (SUV) based on quantitative score normalized to liver (SUV vessel max/liver mean)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Daikeler, Prof. Dr. MD, Principal Investigator — Department of Rheumatology, University Hospital Basel
Locations (1):
- Department of Rheumatology, University Hospital Basel, Basel, Switzerland

REFERENCES:
- [Background] Stone JH, Tuckwell K, Dimonaco S, Klearman M, Aringer M, Blockmans D, Brouwer E, Cid MC, Dasgupta B, Rech J, Salvarani C, Schett G, Schulze-Koops H, Spiera R, Unizony SH, Collinson N. Trial of Tocilizumab in Giant-Cell Arteritis. N Engl J Med. 2017 Jul 27;377(4):317-328. doi: 10.1056/NEJMoa1613849. PMID 28745999
- [Background] Restuccia G, Boiardi L, Cavazza A, Catanoso M, Macchioni P, Muratore F, Cimino L, Aldigeri R, Crescentini F, Pipitone N, Salvarani C. Flares in Biopsy-Proven Giant Cell Arteritis in Northern Italy: Characteristics and Predictors in a Long-Term Follow-Up Study. Medicine (Baltimore). 2016 May;95(19):e3524. doi: 10.1097/MD.0000000000003524. PMID 27175649
- [Background] Kermani TA, Sreih AG, Cuthbertson D, Carette S, Hoffman GS, Khalidi NA, Koening CL, Langford CA, McAlear CA, Monach PA, Moreland L, Pagnoux C, Seo P, Warrington KJ, Ytterberg SR, Merkel PA; Vasculitis Clinical Research Consortium. Evaluation of damage in giant cell arteritis. Rheumatology (Oxford). 2018 Feb 1;57(2):322-328. doi: 10.1093/rheumatology/kex397. PMID 29112740
- [Background] Quinn KA, Ahlman MA, Malayeri AA, Marko J, Civelek AC, Rosenblum JS, Bagheri AA, Merkel PA, Novakovich E, Grayson PC. Comparison of magnetic resonance angiography and 18F-fluorodeoxyglucose positron emission tomography in large-vessel vasculitis. Ann Rheum Dis. 2018 Aug;77(8):1165-1171. doi: 10.1136/annrheumdis-2018-213102. Epub 2018 Apr 17. PMID 29666047
- [Background] Dejaco C, Ramiro S, Duftner C, Besson FL, Bley TA, Blockmans D, Brouwer E, Cimmino MA, Clark E, Dasgupta B, Diamantopoulos AP, Direskeneli H, Iagnocco A, Klink T, Neill L, Ponte C, Salvarani C, Slart RHJA, Whitlock M, Schmidt WA. EULAR recommendations for the use of imaging in large vessel vasculitis in clinical practice. Ann Rheum Dis. 2018 May;77(5):636-643. doi: 10.1136/annrheumdis-2017-212649. Epub 2018 Jan 22. PMID 29358285
- [Background] Attenberger UI, Liu J, Riffel P, Budjan J, Grimm R, Block KT, Schoenberg SO, Wang X, Hausmann D. Quantitative Perfusion Analysis of the Rectum Using Golden-Angle Radial Sparse Parallel Magnetic Resonance Imaging: Initial Experience and Comparison to Time-Resolved Angiography With Interleaved Stochastic Trajectories. Invest Radiol. 2017 Dec;52(12):715-724. doi: 10.1097/RLI.0000000000000397. PMID 28622248
- [Background] Riffel P, Zoellner FG, Budjan J, Grimm R, Block TK, Schoenberg SO, Hausmann D. "One-Stop Shop": Free-Breathing Dynamic Contrast-Enhanced Magnetic Resonance Imaging of the Kidney Using Iterative Reconstruction and Continuous Golden-Angle Radial Sampling. Invest Radiol. 2016 Nov;51(11):714-719. doi: 10.1097/RLI.0000000000000299. PMID 27299581
- [Background] Parikh N, Ream JM, Zhang HC, Block KT, Chandarana H, Rosenkrantz AB. Performance of simultaneous high temporal resolution quantitative perfusion imaging of bladder tumors and conventional multi-phase urography using a novel free-breathing continuously acquired radial compressed-sensing MRI sequence. Magn Reson Imaging. 2016 Jun;34(5):694-8. doi: 10.1016/j.mri.2015.12.033. Epub 2015 Dec 29. PMID 26740058
- [Background] Rosenkrantz AB, Geppert C, Grimm R, Block TK, Glielmi C, Feng L, Otazo R, Ream JM, Romolo MM, Taneja SS, Sodickson DK, Chandarana H. Dynamic contrast-enhanced MRI of the prostate with high spatiotemporal resolution using compressed sensing, parallel imaging, and continuous golden-angle radial sampling: preliminary experience. J Magn Reson Imaging. 2015 May;41(5):1365-73. doi: 10.1002/jmri.24661. Epub 2014 May 16. PMID 24833417
- [Background] Reichenbach S, Adler S, Bonel H, Cullmann JL, Kuchen S, Butikofer L, Seitz M, Villiger PM. Magnetic resonance angiography in giant cell arteritis: results of a randomized controlled trial of tocilizumab in giant cell arteritis. Rheumatology (Oxford). 2018 Jun 1;57(6):982-986. doi: 10.1093/rheumatology/key015. PMID 29529280
- [Background] Blockmans D, de Ceuninck L, Vanderschueren S, Knockaert D, Mortelmans L, Bobbaers H. Repetitive 18F-fluorodeoxyglucose positron emission tomography in giant cell arteritis: a prospective study of 35 patients. Arthritis Rheum. 2006 Feb 15;55(1):131-7. doi: 10.1002/art.21699. PMID 16463425
- [Background] Martinez-Rodriguez I, Jimenez-Alonso M, Quirce R, Jimenez-Bonilla J, Martinez-Amador N, De Arcocha-Torres M, Loricera J, Blanco R, Gonzalez-Gay MA, Banzo I. 18F-FDG PET/CT in the follow-up of large-vessel vasculitis: A study of 37 consecutive patients. Semin Arthritis Rheum. 2018 Feb;47(4):530-537. doi: 10.1016/j.semarthrit.2017.08.009. Epub 2017 Aug 31. PMID 28967430
- [Background] Grayson PC, Alehashemi S, Bagheri AA, Civelek AC, Cupps TR, Kaplan MJ, Malayeri AA, Merkel PA, Novakovich E, Bluemke DA, Ahlman MA. 18 F-Fluorodeoxyglucose-Positron Emission Tomography As an Imaging Biomarker in a Prospective, Longitudinal Cohort of Patients With Large Vessel Vasculitis. Arthritis Rheumatol. 2018 Mar;70(3):439-449. doi: 10.1002/art.40379. Epub 2018 Feb 6. PMID 29145713
- [Background] Imfeld S, Rottenburger C, Schegk E, Aschwanden M, Juengling F, Staub D, Recher M, Kyburz D, Berger CT, Daikeler T. [18F]FDG positron emission tomography in patients presenting with suspicion of giant cell arteritis-lessons from a vasculitis clinic. Eur Heart J Cardiovasc Imaging. 2018 Aug 1;19(8):933-940. doi: 10.1093/ehjci/jex259. PMID 29126277
- [Background] Ironi G, Tombetti E, Napolitano A, Campolongo M, Fallanca F, Incerti E, Picchio M, Dagna L, Manfredi AA, Gianolli L, Del Maschio A, De Cobelli F. Diffusion-Weighted Magnetic Resonance Imaging Detects Vessel Wall Inflammation in Patients With Giant Cell Arteritis. JACC Cardiovasc Imaging. 2018 Dec;11(12):1879-1882. doi: 10.1016/j.jcmg.2018.06.015. Epub 2018 Aug 15. No abstract available. PMID 30121275